CLINICAL TRIAL: NCT03536000
Title: Evaluation of Fetal Cardiac Function With aCMQ-STRAIN: Normality Curve and Comparison to Fetus With Cardiac Disfunction Risk Factors
Brief Title: Fetal Cardiac Function Evaluation With aCMQ-Strain Fetal (STRAIN)
Acronym: STRAIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CMQ-2017-99
Record Dates: First submitted 2018-05-03; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Fetal Cardiac Disorder
Keywords: Cardiac function; Fetal; Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy women: * 200 Pregnant women
  * Over 18 years
  * Healthy
  * With the ability to understand and sign the informed Consent
  * With the ability to attend the established controls
  * Fetal echocardiography using the aCMQ-Strain method (Automated Cardiac Motion Quantification) at 24, 28, 32 and 36 weeks of gestation
  Interventions: Diagnostic Test: Fetal echocardiography using the aCMQ-Strain method
- Intrauterine Growth restriction: * Pregnant women
  * Over 18 years
  * Intrauterine Growth Reestriction(IUGR): fetuses with percentile Growth <p3 or <p10 with vascular Doppler alteration.
  * With the ability to understand and sign the informed Consent
  * With the ability to attend the established controls
  * Fetal echocardiography using the aCMQ-Strain method (Automated Cardiac Motion Quantification) at 24, 28, 32 and 36 weeks of gestation
  Interventions: Diagnostic Test: Fetal echocardiography using the aCMQ-Strain method
- Preeclampsia: * Pregnant women
  * Over 18 years
  * Preeclampsia: elevated blood pressure + Ratio Prot/Creatinin in urine> 30 mg / mmol creatinin
  * With the ability to understand and sign the informed Consent
  * With the ability to attend the established controls
  * Fetal echocardiography using the aCMQ-Strain method (Automated Cardiac Motion Quantification) at 24, 28, 32 and 36 weeks of gestation
  Interventions: Diagnostic Test: Fetal echocardiography using the aCMQ-Strain method
- Diabetes Mellitus type 1: * Pregnant women
  * Over 18 years
  * Diabetes mellitus type1
  * With the ability to understand and sign the informed Consent
  * With the ability to attend the established controls
  * Fetal echocardiography using the aCMQ-Strain method (Automated Cardiac Motion Quantification) at 24, 28, 32 and 36 weeks of gestation
  Interventions: Diagnostic Test: Fetal echocardiography using the aCMQ-Strain method

INTERVENTIONS:
Diagnostic Test: Fetal echocardiography using the aCMQ-Strain method — Fetal echocardiography using the aCMQ-Strain method (Automated Cardiac Motion Quantification) at 24, 28, 32 and 36 weeks of gestation

SUMMARY:
To assess whether the aCQM-Strain ultrasound method allows a good analysis of fetal cardiac function. Establish normality parameters and compare it with fetuses with risk factors of cardiac dysfunction.

DETAILED DESCRIPTION:
National unicentric observational study of follow-up study of a cohort. It has been decided to conduct a study of consecutive cases, including all patients who meet the inclusion criteria during the time of the study.

Until now, there has not been an easy and convenient method to determine fetal cardiac function. Recently a new Software (Automated Cardiac Motion Quantification aCMQ) has been developed, and it seems that allows an easier analysis of this one.

This study aims to analyze fetal heart function with the Strain method in healthy patients and then compare it with fetuses with risk factors for cardiac dysfunction.

Initially, healthy pregnant patients who agree to participate in the study will be cited, after signing the informed consent, in order to evaluate the normal fetal cardiac function and see how it is modified in the different weeks of gestation.

To do this, a fetal echocardiography will be performed by the investigators at week 24, 28, 32 and 36 of pregnancy, using the aCMQ-Strain method.

Once the investigators have established normality curves, fetuses with risk factors for cardiac dysfunction of women who agree to participate in the study will be analyzed. For this purpose, a fetal echocardiography at week 24, 28, 32 and 36 of gestation, using the aCMQ-Strain method will be performed.

All tests will be carried out in the same study center and will be carried out by independent scouts.The data obtained in each test will be collected in an anonymized database for further study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Pregnant women> 20 weeks gestation
* Understand and accept the study procedures and sign an informed consent.

Exclusion Criteria:

* Not being able to understand the nature of the study and / or the procedures to be followed.
* Not signing informed consent
* Under 18 years of age
* Not pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those healthy pregnant women who come to our hospital to perform the morphological ultrasound of the 2nd trimester, or pregnant women with pregestational diabetes, or with a diagnosis of intrauterine growth restriction and / or preeclampsia will be invited to participate in the study. For this, the Participant Information sheet in the study will be provided and the Informed Consent will be signed.
  Those patients who wish to participate in the study will be cited for the performance of an echocardiography using the aCMQ-Strain method at week 24, 28, 32 and 36 of gestation.
  All the tests will be carried out in the same study center and will be carried out by independent scouts.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-05-28 (Estimated); Primary Completion 2019-04-11 (Estimated); Study Completion 2019-09-11 (Estimated)

PRIMARY OUTCOMES:
Changes in the shortening of cardiac fibers during cardiac cycle | At 24, 28, 32 and 36 weeks of gestation
  Fetal echocardiography using the aCMQ-Strain method (Automated Cardiac Motion Quantification)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa LLurba, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Mieghem T. Re: Descriptive analysis of different phenotypes of cardiac remodeling in fetal growth restriction. M. Rodriguez-Lopez, M. Cruz-Lemini, B. Valenzuela-Alcaraz, L. Garcia-Otero, M. Sitges, B. Bijnens, E. Gratacos and F. Crispi. Ultrasound Obstet Gynecol 2017; 50: 207-214. Ultrasound Obstet Gynecol. 2017 Aug;50(2):154. doi: 10.1002/uog.17541. No abstract available. PMID 28782233
- [Background] Crispi F, Gratacos E. Fetal cardiac function: technical considerations and potential research and clinical applications. Fetal Diagn Ther. 2012;32(1-2):47-64. doi: 10.1159/000338003. Epub 2012 May 17. PMID 22614129
- [Background] Comas M, Crispi F, Cruz-Martinez R, Martinez JM, Figueras F, Gratacos E. Usefulness of myocardial tissue Doppler vs conventional echocardiography in the evaluation of cardiac dysfunction in early-onset intrauterine growth restriction. Am J Obstet Gynecol. 2010 Jul;203(1):45.e1-7. doi: 10.1016/j.ajog.2010.02.044. Epub 2010 May 10. PMID 20451892